CLINICAL TRIAL: NCT01035411
Title: An Open-label, Single-centre, 3-way Single Dose Crossover Study to Assess the Relative Bioavailability After Oral Administration of a Tablet Variant of AZD9668 Compared to AZD9668 Tablets and to Further Investigate the Safety and Tolerability of AZD9668 in Healthy Subjects
Brief Title: AZD9668 Relative Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D0520C00007
Record Dates: First submitted 2009-12-14; First posted 2009-12-18 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD9668 2X30mg tablet
  Interventions: Drug: AZD9668

INTERVENTIONS:
Drug: AZD9668 — 2 x 30 mg batch DLE494
Drug: AZD9668 — 2 x 30 mg batch DLF497
Drug: AZD9668 — 2 x 30 mg tablet variant 1

SUMMARY:
This clinical study will aid future formulation development and optimisation of AZD9668 tablets by evaluating possible effects of minor changes to the formulation and process on the rate and extent of absorption.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* female subjects may be of non-child bearing potential (i.e. post menopausal or surgically sterile) or of child bearing potential
* Body mass index (BMI) ≥18.0 and ≤30.0 kg/m2 calculated from height and weight at the screening visit; minimum weight 50 kg.
* Clinically normal physical and laboratory findings as judged by the investigator, including negative test results for drug-of-abuse, alcohol, cotinine and negative test results for Hepatitis B surface antigen, antibodies to Hepatitis C virus and antibodies to HIV-1/2 at the screening visit
* Be a none smoker or ex-smoker who has stopped smoking for >6 months prior to visit 2 (pre-entry)

Exclusion Criteria:

* Any clinically significant disease or disorder (eg infections/viral disease, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment), which in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the absorption, distribution, metabolism and excretion of drugs.
* Any clinically relevant abnormal findings in physical examination, vital signs, clinical chemistry, haematology, urinalysis, which, in the opinion of the investigator, may put the subject at risk because of his/her participation in the study
* Any ECG abnormality (including cardiac arrhythmia) which in the opinion of the investigator may put the subject at risk

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (Frel): to assess the relative systemic bioavailability after oral administration of a tablet variant of AZD9668 compared to AZD9668 tablets. | Frequent sampling occasions during the study

SECONDARY OUTCOMES:
Safety variables (adverse events, vital signs, haematology, clinical chemistry, urinalysis and 12-lead ECG) | Frequent sampling occasions during the study

CONTACTS AND LOCATIONS:
Overall Officials: Emma Harrop, Study Director — AstraZeneca R&D; Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany